CLINICAL TRIAL: NCT01515020
Title: A Randomized, Multicenter Trial of Daptomycin Versus Vancomycin in the Treatment of Nosocomial or Healthcare-associated Methicillin-resistant Staphylococcus Aureus Bacteremia
Brief Title: Daptomycin Versus Vancomycin in the Treatment of Nosocomial or Healthcare-associated MRSA Bacteremia
Acronym: DAVASAB
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P100110; AOM10082 (Other: French Ministry)
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Nosocomial Infection; Healthcare-associated Infection
Keywords: bacteremia; meticillin-resistant Staphylococcus aureus; nosocomial infection; healthcare-associated infection; rapid molecular diagnostic test
MeSH Terms: conditions — Cross Infection; Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- vancomycin monotherapy (Active Comparator): vancomycin monotherapy: standard therapy
  Interventions: Drug: vancomycin monotherapy
- daptomycin monotherapy (Experimental): daptomycin monotherapy: experimental therapy
  Interventions: Drug: daptomycin monotherapy

INTERVENTIONS:
Drug: vancomycin monotherapy — intravenous therapy by vancomycin
  Other Names: intravenous therapy
  Arms: vancomycin monotherapy
Drug: daptomycin monotherapy — intravenous therapy by daptomycin
  Other Names: intravenous therapy
  Arms: daptomycin monotherapy

SUMMARY:
Hypothesis: The use of daptomycin to treat nosocomial or healthcare-associated bacteremia due to methicillin-resistant S. aureus (MRSA) would increase the proportion of patients whose blood cultures are sterilized after 72 hours by 15% relative to vancomycin and would improve treatment safety.

Hypothesis: for MRSA nosocomial or healthcare related bacteriemia treatment, the use of daptomycin versus vancomycin would increase by 15% the proportion of patients with sterilized blood cultures at 72 hours and would increase the treatment safety.

Primary objective: To study the efficacy of daptomycin compared to vancomycin on the sterilization of blood cultures after 72 hours of therapy.

DETAILED DESCRIPTION:
Introduction: Nosocomial and/or healthcare-associated Staphylococcus aureus infections are common, serious conditions. S. aureus accounts for about 20% of cases of nosocomial bacteremia, and is associated with a mortality of 20-40%. This severity is due to the virulence of the bacterium, and the age and comorbidity of the patients in whom the infection occurs. First-line therapy is based on vancomycin, because the prevalence of methicillin resistance in S. aureus (~20%) is still high in the hospital environment. However the bactericidal activity of this drug is slow and it causes dose-dependent nephrotoxicity. The persistence of positive blood cultures after 72 hours, a parameter which in itself is predictive of the infection having a complicated clinical course, is seen in about 35% of patients receiving vancomycin therapy.

Hypothesis: The use of daptomycin to treat nosocomial or healthcare-associated bacteremia due to methicillin-resistant S. aureus (MRSA) would increase the proportion of patients whose blood cultures are sterilized after 72 hours by 15% relative to vancomycin and would improve treatment safety.

Primary objective: To study the efficacy of daptomycin compared to vancomycin on the sterilization of blood cultures after 72 hours of therapy.

Secondary objectives: Clinical cure at D14 and D28; relapse-free clinical and bacteriological cure at D90; mortality at D14, D28 and D90; treatment duration (in days) before sterilization of blood cultures; side effects occurrence during treatment, renal insufficiency; peripheral vein toxicity requiring placement of a central venous catheter; side effects requiring changes to the study treatment ; duration of hospitalization for bacteremia; increase of at least 2 dilutions in the minimal inhibitory concentration (MIC) of daptomycin and/or vancomycin between the first and last clinical isolates of S. aureus.

Methodology: A prospective, multicenter, randomized, open-label study to compare daptomycin monotherapy to vancomycin monotherapy. Patients will be randomized if they have a nosocomial or healthcare-associated infection, a blood culture positive for Gram-positive cocci in clusters, and a rapid molecular diagnostic test(GENEXPERT) that confirm the presence of methicillin-resistant S. aureus. Daptomycin will be given once daily in monotherapy (10 mg/kg as a single infusion over 30 minutes into a peripheral vein). Standard therapy is vancomycin in monotherapy given by intermittent or continuous infusion so as to obtain trough concentrations of 15-20 mg/L or plateau concentrations of 20-25 mg/L, respectively. The treatment duration for bacteremia in both arms is 14 days of intravenous therapy for uncomplicated bacteremias and 28 days of intravenous therapy for complicated bacteremias, defined by persistent fever or positive blood cultures after 72 h of the study treatment, secondary septic localizations existing at enrollment, or presence of foreign material without signs of infection.

The duration of the treatment of the study can be reduced if the patients answer the following criteria:

Uncomplicated bacteremia: 10 days of treatment instead of 14 days if:

* 2 sterilization of blood cultures
* Patient clinically cured
* Visit J14 realized in the center

Complicated bacteremia: 21 days of treatment instead of 28 days if:

* 2 sterilization of blood cultures
* Patient clinically cured
* Visit J28 realized in the center

In every case, no oral relay has to substitute itself for the possible reduction of the duration of the treatment of the study.

A blinded study design was not selected because the two treatments are administered very differently, due to the invasive nature of continuous infusion pumps, and because the primary objective concerns a microbiological outcome.

Patient management and clinical monitoring will comply with usual good clinical practice for these patients. Visits on D14, D28 and D90 will be necessary. Laboratory monitoring will comprise daily blood cultures until sterile cultures are obtained on 2 consecutive days; full blood count (FBC), serum creatine, CPK before treatment, on D3, D7, D10 and D14 and, for patients receiving 28 days of treatment, D21 and D28. Where myalgia with elevation of creatine phosphokinase (CPK) > 5 N, or isolated elevation of CPK > 10 N occurs, treatment with daptomycin will be discontinued and clinical and laboratory-based monitoring will be maintained until normalization.

Number of subjects required: After 72 hours of vancomycin therapy, blood cultures are still positive in about 35% of patients. The objective is to show the superiority of daptomycin in the sterilization of blood cultures after 72 hours, by a margin of 15% (80% versus 65%). With a power of 80% and a type I error rate of 5%, and addition of 10% to allow for unevaluable outcomes and death before 72 hours, the number of subjects required in each arm is 166 (total = 332 patients).

Study logistics: Duration of the study: 2 years; Enrollment period: 21 months; Duration of each patient's participation: 3 months; Number of participating study sites: 15. Study sites were chosen on the basis of the blood culture system used, of there having been > 10 methicillin-resistant S. aureus blood cultures in 2009 and the possibility of setting up rapid diagnosis for the trial.

A two-person team consisting of a bacteriologist and a clinician will be responsible for [screening], [enrollment] [and] [randomization] at [each] study site.

Mean number of patients enrolled per month per site: 1-5.

ELIGIBILITY:
INCLUSION CRITERIA :

* Patients with nosocomial and/or healthcare-associated bacteremia with Gram-positive cocci in clusters
* Confirmed to be meticillin-resistant S. aureus using a GeneXpert rapid molecular test
* Aged 18 years or older
* Who have given their written consent when this is possible or someone from his/her family, or if not possible, emergency inclusion
* Who can receive follow-up for the entire duration of the study, i.e. 90 days

EXCLUSION CRITERIA :

* Known allergy to vancomycin or daptomycin
* Women who are pregnant or breast-feeding
* Patients who have received vancomycin treatment for more than 48 hours between the diagnostic blood culture and randomization
* Specific sites of infection: pneumonia, meningitis, brain abscess, osteitis, polymicrobial infection
* Life expectancy considered to be less than 72 hours
* Severe hepatic impairment (Child C)
* Short-term intravascular catheters which cannot be removed immediately

EXCLUSION CRITERIA between D1 and D5 inclusive :

* Specific sites of infection: osteitis diagnosed between D1 and D5 inclusive
* Permanent foreign material infection (endovascular stents, replacement heart valves or joints, pace maker etc.) which cannot be removed within 36 hours of the first dose of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Rates of sterilization of blood cultures after 72 hours of therapy | 72 hours
  To study the efficacy of daptomycin compared to vancomycin on the sterilization of blood cultures after 72 hours of therapy.

SECONDARY OUTCOMES:
Clinical cure at D14 | 14 days
  Clinical cure at D14
Clinical cure at D28 | 28 days
  Clinical cure at D28
relapse-free clinical and bacteriological cure at D90 | 90 days
  relapse-free clinical and bacteriological cure at D90
treatment duration (in days) before sterilization of blood cultures | 28 days
  treatment duration (in days) before sterilization of blood cultures
side effects occurrence during treatment | 28 days
  side effects occurrence during treatment
renal insufficiency | 90 days
  renal insufficiency
peripheral vein toxicity requiring placement of a central venous catheter | 28 days
  peripheral vein toxicity requiring placement of a central venous catheter
side effects requiring changes to the study treatment | 28 days
  side effects requiring changes to the study treatment
duration of hospitalization for bacteremia | 90 days
  duration of hospitalization for bacteremia
increase of at least 2 dilutions in the MIC of daptomycin and/or vancomycin between the first and last clinical isolates of S. aureus | 28 days
  increase of at least 2 dilutions in the MIC of daptomycin and/or vancomycin between the first and last clinical isolates of S. aureus

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FANTIN, Pr, Principal Investigator — APHP
Locations (1):
- Hopital Beaujon, Clichy, France